CLINICAL TRIAL: NCT00593307
Title: The Effects of Low and High Glycemic Index Foods and Protein on Glycemic Response and Hunger
Brief Title: The Breakfast Study
Acronym: Breakfast
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Temple University (Other)
Collaborators: International Life Sciences Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 10917; ILSI
Record Dates: First submitted 2008-01-03; First posted 2008-01-15 (Estimated); Last update posted 2013-07-01 (Estimated); Status verified 2008-01

CONDITIONS: Glycemic Response; Hunger
Keywords: glycemic response; hunger

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Low GI (Experimental): low GI breakfast
  Interventions: Other: Low GI
- Low GI -low carb (Experimental): Low GI and Low carb breakfast
  Interventions: Other: Low GI Low Carb
- High GI (Experimental): High GI breakfast
  Interventions: Other: high GI
- High GI Low Carb (Experimental): high GI low carb breakfast
  Interventions: Other: High GI Low carb

INTERVENTIONS:
Other: high GI — high GI and high carb breakfast
  Arms: High GI
Other: Low GI — low GI, high carb breakfast
  Arms: Low GI
Other: Low GI Low Carb — low GI low carb breakfast
  Arms: Low GI -low carb
Other: High GI Low carb — high GI low carb breakfast
  Arms: High GI Low Carb

SUMMARY:
The overall objective is to investigate the effects of low and high glycemic index (GI) meals varying in protein content on plasma glucose and insulin response, subjective ratings of hunger, and subsequent food intake in twenty healthy, sedentary, overweight and obese men and women between the ages of 21-65.

DETAILED DESCRIPTION:
Each individual will participate separately in four testing sessions. Each testing session will last for approximately 5 hours and will be separated by a minimum of one week. Participants will arrive at the Temple University GCRC or CORE at either 7:30 a.m. or 8:30 a.m. after an overnight fast (10-12 hours) to ensure that all participants are in the same metabolic state. Upon arrival the experimenter will ask participants to complete a pre-session questionnaire and rate their feelings of hunger and satiety on a visual analog scale (VAS). An indwelling catheter will be inserted in an antecubital vein by the study nurse and a baseline blood sample will be obtained for measurement of glucose and insulin concentrations. Glucose will be measured by the glucose oxidase method using a glucose analyzer and insulin will be measured by radioimmunoassay.

One of four isocaloric meals (see example below), varying in macronutrient content and GI value of foods, will be administered in random order at either 8:00 a.m. or 9:00 a.m. Energy density will be controlled. The meal and 8 ounces of water will be consumed within fifteen minutes. A short visual analog questionnaire will be distributed at the conclusion of the meal to rate the meal consumed. Blood samples will be taken 15 minutes after food consumption and at 30 minute intervals (i.e., 30, 60, 90, 120, 150, 180, 210, and 240 minutes) over four hours following administration of the meal. Four milliliters of blood will be collected at each time point (via indwelling catheter), resulting in a total of 40 milliliters of blood collected at each study session and 160 milliliters (i.e., 40 ml x 4 testing sessions) within an 8 week time period. Participants will be asked to rate their feelings of hunger at these time points. Following the last blood sample, participants will be given the opportunity to consume food ad libitum from a buffet style lunch. Based on known serving sizes and measurements of unconsumed food, the amount of food eaten and its associated energy content will be determined.

ELIGIBILITY:
Inclusion Criteria:

* Men and women between the ages of 21-65 with a BMI of 25-40(kg/m2)

Exclusion Criteria:

* Individuals who are currently dieting or restricting food intake and who report pre-existing health afflictions such as diabetes, use of prescription medications, use of appetite suppressants, or regular tobacco use will be excluded from the study as they may affect appetite or impact the dependent measures of this study.

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2006-01; Primary Completion 2008-06 (Actual); Study Completion 2008-06 (Actual)

PRIMARY OUTCOMES:
To compare the effects of breakfast meals containing low GI and high GI foods on glucose and insulin responses | post

SECONDARY OUTCOMES:
To examine the effects of low and high GI meals on subjective ratings of hunger and subsequent food intake | post
To compare the effects of high protein meals containing either low or high GI foods with high carbohydrate meals containing either low or high HI food on glucose and insulin response, subjective ratings of hunger, and subsequent food intake. | post

CONTACTS AND LOCATIONS:
Overall Officials: Gary D Foster, PhD, Principal Investigator — Temple University - Center for Obesity Research and Education
Locations (1):
- Temple University - Center for Obesity Research and Education, Philadelphia, Pennsylvania, United States